CLINICAL TRIAL: NCT03030560
Title: Effect of Intravenous Lidocaine Infusion on Long Term Postoperative Pain After Spinal Fusion Surgery
Brief Title: Longterm Postoperative Analgesia, Intravenous Lidocaine Infusion
Acronym: Lidocaine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abdelrady S Ibrahim, MD (Other)
Responsible Party: Sponsor-Investigator, Abdelrady S Ibrahim, MD, Assistant professor of anesthesia and ICU, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB0000871239
Record Dates: First submitted 2017-01-22; First posted 2017-01-25 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine group (Active Comparator): Patients will receive lidocaine infusion.
  Interventions: Drug: Lidocaine
- Control group (Placebo Comparator): Patients will receive 0.9% Sodium-chloride infusion infusion
  Interventions: Drug: 0.9% Sodium-chloride

INTERVENTIONS:
Drug: Lidocaine — patients (n = 20) will receive a loading dose of lidocaine 2 mg ̸ kg slowly IV just before induction of anesthesia, then the lidocaine infusion started at a rate of 3 mg ̸ kg/h, and continued until the end of the operation.
  Other Names: Xylocaine
  Arms: Lidocaine group
Drug: 0.9% Sodium-chloride — patients (n = 20) will receive an equal volume of 0.9% saline (both the loading and the infusion), the infusion will be initiated at the time of induction of anesthesia and continued until the end of the operation.
  Other Names: Normal saline
  Arms: Control group

SUMMARY:
Spinal fusion is a painful surgery, and control of postoperative pain is difficult. Several studies have indicated that appropriate pain treatment protocols reduce postoperative morbidity, improve the results of the surgery, and decrease hospital costs

DETAILED DESCRIPTION:
Forty four patients were randomly allocated into two groups of equal size to receive either lidocaine infusion (Lidocaine group) or 0.9% sodium chloride infusion (Control group).

Randomization: was performed using Lidocaine group and Control group registers, which was placed in sealed envelopes prior to study initiation and opened prior to anesthesia by a physician who prepared the intravenous solution and identified it with the patient number, according to the envelope drawn. The solution was handed to another physician, blind to the prepared solutions' content, who was responsible for the anesthesia. The solution volume was equal. The responsible investigator was remained blind to the chosen group until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years American Society of Anesthesiologists 1-3 status Patients undergoing spinal fusion or fixation

Exclusion Criteria:

1. Previous spinal fusion surgery.
2. Morbid obesity (BMI > 40)
3. Diagnosis of spinal metastatic cancer
4. Allergy to an amide local anesthetic or morphine sulfate
5. History of renal dysfunction, liver dysfunction or congestive heart failure
6. History of substance abuse disorder.
7. Chronic opioid use.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
numerical rating scale (NRS), pain score. | Postoperative 3 months
  Postoperative numerical rating scale (NRS), pain score.

SECONDARY OUTCOMES:
opioid consumption. | Postoperative 24 h
  Postoperative opioid consumption.
Serum cortisol. | Postoperative 24 h
  Serum cortisol level.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed G Abdelraheem, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Oliveira CM, Issy AM, Sakata RK. Intraoperative intravenous lidocaine. Rev Bras Anestesiol. 2010 May-Jun;60(3):325-33. doi: 10.1016/S0034-7094(10)70041-6. PMID 20682165